CLINICAL TRIAL: NCT04127968
Title: Efficacy and Safety of Vitamin A Treatment for Children With Sepsis: a Randomized Placebo-controlled Clinical Trial
Brief Title: Efficacy and Safety of Vitamin A Treatment for Children With Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, MD, PhD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1010
Record Dates: First submitted 2019-10-12; First posted 2019-10-16 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Vitamin A Deficiency; Pediatric; Sepsis
MeSH Terms: conditions — Vitamin A Deficiency; Sepsis | interventions — Vitamin A; Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Septic children with vitamin A deficiency who will receive vitamin A supplementation.
  Interventions: Drug: Vitamin A
- control group (Placebo Comparator): Septic children with vitamin A deficiency who will receive placebo.
  Interventions: Drug: Oil

INTERVENTIONS:
Drug: Vitamin A — Children in intervention group will receive 50,000 IU vitamin A after being randomized.
  Arms: intervention group
Drug: Oil — Children in control group will receive equal volume of oil.
  Arms: control group

SUMMARY:
The prevalence of vitamin A deficiency was found high in children with sepsis. Whether those patients will benefit from the vitamin A supplementation is unknown.

DETAILED DESCRIPTION:
It was reported that the prevalence of vitamin A deficiency was highly as 58% in critically ill children with sepsis. However, whether those patients will benefit from the vitamin A supplementation is unknown. We design an randomized, double-blind, placebo-controlled, multi-center trial to investigate the effect of vitamin A supplementation on the outcome of critically ill children with sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. age < 18 years,
2. Expected to stay in the ICU for 48 hours or more,
3. Vitamin A deficiency (VA < 0.2 mg/L)

Exclusion Criteria:

1. Severely impaired gastrointestinal function
2. Premature infants and low birth weight (LBW) infants
3. Condition of underlying organ dysfunction
4. Having received chemotherapy or radiotherapy
5. Hematological malignancies
6. Primary or acquired immunodeficiency

Ages: 0 Months to 192 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
length of hospital stay | 2 years
  The length of hospital stay will be measured by days

SECONDARY OUTCOMES:
hospital mortality | 2 years
  Hospital mortality will be record as ratio

REFERENCES:
- [Derived] Fu Q, Liu M, Zhang X, Fu J, Zhang G, Ji Y, Chen S. A randomized controlled trial on the efficacy and safety of vitamin A supplementation in children with sepsis. Front Pediatr. 2025 Aug 6;13:1579006. doi: 10.3389/fped.2025.1579006. eCollection 2025. PMID 40843069